CLINICAL TRIAL: NCT03457402
Title: Feasibility of Shaping Tolerance for Delayed Rewards in Impulsive 3-6 Year Olds
Brief Title: Shaping Tolerance for Delayed Rewards
Acronym: DelTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 921404; R03HD087091-01A1 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Impulsivity
Keywords: delay discounting; shaping
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two possible groups.
  Group 1: Treatment; this group begins 6-week training with the self-control shaping application immediately after baseline.
  Group 2: Wait-list Control; After baseline, this group waits for 6-weeks before completing another pre-training assessment and then starts the 6-week training with the self-control application.
Who Masked: Outcomes Assessor
Masking Description: Care Providers are told about the two possible groups during the Consent and will be aware of their child's assignment in terms of whether the child begins treatment immediately after baseline or has to wait 6 weeks prior to treatment.
  Members of the research team who are designated as video coders for the Effortful Control tasks will be blind to the group assignment of the participants in the video recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the Experimental arm will begin the Shaping Delay Tolerance behavioral intervention immediately after baseline, and this training will last for about 6 weeks.
  Interventions: Behavioral: Shaping Delay Tolerance
- Wait-list Control (Active Comparator): After baseline, participants in the Wait-list Control arm will wait for about 6-weeks before entering the pre-treatment phase, which is a repeat of effortful control assessments and behavior questionnaires, and then they will begin training for with the Shaping Delay Tolerance behavioral intervention.
  Interventions: Behavioral: Shaping Delay Tolerance

INTERVENTIONS:
Behavioral: Shaping Delay Tolerance — Participants will be introduced to an adaptive tablet-based application that asks the child to choose between two options: 1) a shorter duration of game play that begins immediately, or 2) a longer duration of game play that begins after a delay. Depending on the child's choices, the application alters the pre-reward delay with the intent of training the child to tolerate longer delays for larger rewards (i.e., more game play). Children may participate in up to 25 approximately 30-minute training sessions over 3-6 weeks.

SUMMARY:
Deficits in self-control are of major public health relevance as they contribute to several negative outcomes for both individuals and society. For children, developing self-control is a critically important step toward success in academic settings and social relationships, yet there are few non-pharmacological approaches that have been successful in increasing self-control. We found in our earlier studies that self-control can be increased in preschool-aged children with high impulsivity by using games in which they practice gradually increasing wait-time for larger, more delayed rewards. We are performing this current study to test if this training to increase self-control can be increased using mobile app technology, with computerized game time being used as a reward.

DETAILED DESCRIPTION:
Problems with self-control are of major public health relevance as they are associated with substance abuse, suicide attempts, lower academic functioning, poor financial planning, and physical and mental health issues that impact both individuals and society. The ability to obtain immediate rewards in our daily lives is increasing due to technological advances from on-line games to Amazon deliveries within 1 hour after placing an order. There are fewer opportunities for children to learn how to wait. For children, developing self-control is a critically important step toward success in academic settings and social relationships, yet there are few non-pharmacological approaches that have been successful in increasing self-control.

Our objective in this current proof-of-concept study is to replicate and extend our earlier finding (Schweitzer & Sulzer-Azaroff, 1988) in which we demonstrated that self-control could be increased in preschool-aged children with high rates of impulsivity by using a "shaping" procedure whereby delays to larger, more delayed rewards were gradually increased. In this study we will aim to show that shaping self-control can be implemented using more sophisticated experimental design and mobile app technology.

A principal goal of this R03 pilot project is to refine the procedural methods to ensure that they are developmentally-appropriate using a well-controlled design and procedures. Our plan is to develop and implement a mobile application ("app"), "Delay Tolerance Application" (DelTA) that administers real-time rewards in a delay discounting procedure, in which the child will choose between an immediate, shorter game playing and a delayed, longer version of playing the same game.

This project will assess the feasibility of delivering the procedure via a mobile app and test if computerized games are effective rewards in a delay discounting context for young children (3-6 years) given that previous methods used immediately consumable rewards (e.g., candy). Positive findings from this proof-of-concept project will support future clinical trial projects to improve self-control and the use of the procedure for other interventions. The app may eventually serve as a targeted, precision intervention for children who exhibit elevated impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-6 years
* Hyperactivity/Impulsivity subscale scores of the ADHD Rating Scale-IV Preschool Version (children 3 to 4 years of age) or the Attention and Behavior Scale (children 5 to 6 years of age) ≥ 90th percentile from either the parent or teacher's responses
* Physically and visually able to use the tablet, as determined by pre-assessment performance
* Children taking psychotropic medication will be included, but must maintain the same medication and dose over the course of the study and for each assessment and exhibit elevated levels of impulsivity based on parent or teacher ratings while medicated.

Exclusion Criteria:

* Children with autism spectrum disorder and/or intellectual disability (by parent or teacher report or the NIH Toolbox Picture Vocabulary Test).

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Indifference point | Up to 6 weeks
  The indifference point on the tablet-task assessment is defined as the delay interval at which the child chooses 50% longer, larger rewards and 50% shorter, smaller rewards. Investigators hypothesize that the shaping group will have greater increases in their indifference points than the waitlist control group.
Percent change in preference for longer, larger (LL) rewards | Up to 6 weeks
  The percentage of trials in which the child selects the longer, larger (LL) reward option during the tablet-task assessment will be recorded. Investigators hypothesize that the shaping group will have greater increases in the percentage of trials for which they choose the LL rewards compared to the waitlist control group.

SECONDARY OUTCOMES:
ADHD-RS-IV Preschool Version and Attention and Behavior Rating Form | Up to 6 weeks
  Parent and teacher ratings regarding the frequency of inattentive and hyperactivity/impulsivity ADHD symptoms. Investigators predict that the shaping group will have better improvement in parent and teacher of ratings of impulsivity than the waitlist control group.
The Preschool Life Skills Questionnaire | Up to 6 weeks
  A 13-item teacher scale that assesses behaviors noted as important to educators in predicting preschool success: instruction following, functional communication, delay tolerance, and friendship skills. Investigators predict the greatest change in the delay tolerance scale in the shaping group compared to the waitlist control.
The Children's Behavior Questionnaire (CBQ) | Up to 6 weeks
  A highly differentiated assessment of temperament in early to middle childhood. Investigators predict the greatest change in the shaping group compared to the waitlist control.
Snack Delay Task | Up to 6 weeks
  An assessment of delay of gratification. In this task, the child is invited to play a game in which he or she is asked to wait for varying intervals (5 seconds, 10 seconds, 20 seconds, 30 seconds) before they can a a parent-approved treat. Behavior is coded for latency to touch and eat the snack (seconds). Investigators predict that the shaping group will have better improvement in delay of gratification in the Snack Delay Task compared to the waitlist control group.
Dinky Toy Task | Up to 6 weeks
  An assessment of effortful control. In this task, the child is asked to look through a prize box containing toys while keeping his hands flat on the table. The child should then select a prize verbally by indicating the name of the toy or providing a description of it. Behavior is coded for latency to choose a prize and whether hands were removed from the designated table mat. Investigators predict that the shaping group will have better improvement in effortful control as measured by the Dinky Toy Task compared to the waitlist control group.
Gift Wrap and Gift Delay Task | Up to 6 weeks
  An assessment of effortful control. In this task, the experimenter shows the child a bag containing a present that still needs to be wrapped. The child is told "try not to look" at the present during the wrapping process, which is completed by the experimenter at a table behind the child's back. The rule is to not peek at the gift. Sixty seconds later, when the experimenter has completed wrapping the gift, she will leave the room to search for a bow while instructing the child not to touch the present. The experimenter returns in 3 minutes, places the bow, and awards the gift. Behavior will be coded for the child's peeking strategy, and his latency to peek at the gift, touch the gift, and leave his seat while the experimenter is away. Investigators predict that the shaping group will have better improvement in effortful control as measured by the Gift Wrap and Gift Delay Task compared to the waitlist control group.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schweitzer, Ph.D., Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

REFERENCES:
- [Background] Schweitzer JB, Sulzer-Azaroff B. Self-control: teaching tolerance for delay in impulsive children. J Exp Anal Behav. 1988 Sep;50(2):173-86. doi: 10.1901/jeab.1988.50-173. PMID 3193054
- [Background] Schweitzer JB, Sulzer-Azaroff B. Self-control in boys with attention deficit hyperactivity disorder: effects of added stimulation and time. J Child Psychol Psychiatry. 1995 May;36(4):671-86. doi: 10.1111/j.1469-7610.1995.tb02321.x. PMID 7650090
- [Background] McGoey KE, DuPaul GJ, Haley E, et al. Parent and teacher ratings of attention-deficit/hyperactivity disorder in preschool: the ADHD Rating Scale-IV Preschool Version. J Psychopathol Behav Assess. 2007;29:269.
- [Background] Dunn LM, Dunn DM. Peabody Picture Vocabulary Test - Fourth Edition (PPVT-4). 2006. Toronto; Pearson: 2006.
- [Background] Hanley GP, Heal NA, Tiger JH, Ingvarsson ET. Evaluation of a class wide teaching program for developing preschool life skills. J Appl Behav Anal. 2007 Summer;40(2):277-300. doi: 10.1901/jaba.2007.57-06. PMID 17624068
- [Background] Rothbart MK, Ahadi SA, Hershey KL, Fisher P. Investigations of temperament at three to seven years: the Children's Behavior Questionnaire. Child Dev. 2001 Sep-Oct;72(5):1394-408. doi: 10.1111/1467-8624.00355. PMID 11699677
- [Background] Putnam SP, Rothbart MK. Development of short and very short forms of the Children's Behavior Questionnaire. J Pers Assess. 2006 Aug;87(1):102-12. doi: 10.1207/s15327752jpa8701_09. PMID 16856791
- [Background] Gagne JR, Van Hulle CA, Aksan N, Essex MJ, Goldsmith HH. Deriving childhood temperament measures from emotion-eliciting behavioral episodes: scale construction and initial validation. Psychol Assess. 2011 Jun;23(2):337-53. doi: 10.1037/a0021746. PMID 21480723
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] Liang K, Zeger S. Longitudinal data analysis using generalized linear models. Biometrika 73:13-22; 1986.